CLINICAL TRIAL: NCT05048446
Title: Physical Activity, Musculoskeletal Disorders, Perception of Emotional Work Well-being and Quality of Life in Professional Musicians
Brief Title: Physical and Work Variables in Professional Musicians
Acronym: SActMWQoLMU
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Other Study IDs: ID0035
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational — Non intervention

SUMMARY:
In professional musicians there are characteristic diseases. In this area there is no preventive culture and many musicians end their professional careers due to ailments and pathologies that cause the abandonment of the profession or they learn to live and play with pain. It is a very demanding profession that requires many hours of training without respecting the necessary rest, which undoubtedly produces fatigue and muscle overload, neurological disorders, etc. Also, the demands to achieve perfection lead to serious work problems.

Given that it is a profession that suffers from pain and psychosomatic alterations and that is often accompanied by emotional alterations due to work demands, it is necessary to know this problem and to what extent it affects the musician to be able to act from different areas and improve his well-being.

The objective is to know specifically the characteristics of professional musicians, their impact variables, both musculoskeletal and emotional, variables related to the workplace and to evaluate their quality of life.

DETAILED DESCRIPTION:
MATERIAL AND METHODS Subjects. Professional orchestral and band musicians between the ages of 18 and 65.

Study design. Descriptive study to be carried out at the University of Valencia. To do this, a survey will be carried out through an online platform. All participants will sign the informed consent and the study will be carried out in compliance with the data confidentiality guidelines. To start the study, the approval of the Ethics Committee of the University of Valencia will be necessary and it will be included in an international registry.

Evaluation. In the first place, the anthropometric data (age, sex, weight, height) and the characteristics of the sample will be taken through an interview designed for this study that will contain questions about the job and instruments they practice. Subsequently, the subjects will fill in the assessment instruments that include the physical activity they perform, the musculoskeletal alterations, workplace harassment, professional burnout, quality of life and anxiety and depression.

Statistic analysis. The variables will be coded and analyzed using the SPSS v.26 program.

ELIGIBILITY:
Inclusion Criteria:

* active professional musicians

Exclusion Criteria:

* non-active or non-practicing professional musicians

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Professional musicians of orchestras and bands
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Physical activity | 1 day
  By Ipaq Short Form. The short form records activity at four levels of intensity: 1) vigorous intensity activity such as aerobics, 2) moderate intensity activity such as leisure riding a bike, 3) walking and 4) sitting.
Musculoskeletal disorders | 1 day
  Will be evaluated by the Nordic questionnaire, this tool is used to detect symptoms musculoskeletal such as pain, discomfort, numbness or tingling. It includes two important sections: The first is choice questions mandatory in which the subject marks the areas of the body where pain occurs; The second section contains related questions on the functional impact of pain symptoms. Also the duration of problem, if it has been evaluated by a health professional and the evolution of pain. This questionnaire does not have a score as such, it does not have a scale to assess it, but rather what, based on the data, the analysis is extracted for each question.

SECONDARY OUTCOMES:
Workplace Harassment | 1 day
  To assess mobbing at work we used the Short-Negative Acts Questionnaire (NAQ). It consists of 9 items of the NAQ. This is a questionnaire that collects typical harassment behaviors, with respect to which the subject must indicate the degree to which they have suffered such behaviors during the last six months. The response scale consists of five alternatives from 1 ("never") to 5 ("daily"). Some examples of the items included are: "Gossip and rumors have spread about me", "I have been the object of offenses about my person or my private life".
Health | 1 day
  The SF-8 questionnaire is structured with eight articles. It is divided into eight subscales (physical functioning, physical role, body pain, general health, vitality, social functioning, emotional role mental and mental health) and two summary components (physical and mental) through which the the results are expressed.
  Scores on the subscales and summary. The components are presented as a mean score of 50. Therefore, scores below 50 points correspond to deviations from normality and indicate a poorer quality of life, while scores above 50 the points represent a better quality of life.
Anxiety and depression | 1 day
  The Golberg scale will be used, a test that orients the diagnosis towards anxiety or depression or both, and discriminates between them and measures their respective intensities. This scale contains 2 subscales with 9 questions each:
  * Anxiety subscale (questions 1-9). If from questions 1-4, a minimum of 2 questions are not answered in the affirmative, the test is not carried out.
  * Depression subscale (questions 10-18). If from questions 10-13, a minimum of 1 questions are not answered in the affirmative, the test is not carried out.
  For its interpretation, the affirmative responses of the Anxiety scale and those of the Depression scale are counted. The cut-off points are 4 or more for the Anxiety subscale and 2 or more for Depression, with scores that are higher the more severe the problem (the maximum possible being 9 in each of the subscales). .
Professional burnout | 1 day
  The Brief Burnout Questionnaire (CBB) will be used. This questionnaire aims to define the Burnout Syndrome or professional burnout syndrome and understand its dimensions. Burnout Syndrome can be defined as the symptoms of exhaustion and emotional exhaustion, the presence of depersonalization and the lack of personal fulfillment that is generated through a process of work stress maintained over time. Three dimensions are contemplated that include the previous factors of Burnout, the development of Burnout Syndrome and the consequences of this Syndrome. The antecedent factors of Burnout include items related to dissatisfaction with the task performed and with the organization in the workplace. The CBB questionnaire consists of 21 items that are evaluated by quantifying the global affectation of the subject by Burnout Syndrome in low, medium or high affectation in each of the three categories mentioned above.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma V E Espí-López, Dr, Principal Investigator — University of Valencia
Locations (2):
- Spain (2):
  - Gemma Espí López, Valencia
  - Gemma Victoria Espí-López, Valencia

IPD SHARING:
Plan to Share IPD: No